CLINICAL TRIAL: NCT04122716
Title: Synergy Effect of the Appetite Hormone GLP-1 (LiragluTide) and Exercise on Maintenance of Weight Loss and Health After a Low Calorie Diet - the S-LiTE Randomized Trial
Brief Title: Combined Effects of GLP-1 Analogue and Exercise on Maintenance of Weight Loss and Health After Very-low Calorie Diet
Acronym: S-LITE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Signe Torekov (Other)
Collaborators: Hvidovre University Hospital (Other); University of Oxford (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Signe Torekov, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U 1111-1173-3104 (UTN); 2015-005585-32 (EudraCT Number); H-16027082 (Other: The Ethical Committee of the Capital Region of Denmark)
Record Dates: First submitted 2018-07-20; First posted 2019-10-10 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: Weight loss maintenance; Immunometabolic health; Exercise intervention; GLP-1 receptor agonist (liraglutide)
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Exercise

STUDY DESIGN:
Intervention Model Description: After 8 weeks of weight loss the participants are randomized to receive a) Liraglutide 3mg/day sc or b) placebo sc or c) Exercise + placebo sc or d) Exercise + Liraglutide 3mg/d sc for 52 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The above-mentioned are masked in terms of Liraglutide/placebo, not in terms of exercise/non-exercise.
  Statistical analysis of primary outcome will be blinded to the assessor.
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (4):
- Liraglutide + exercise (Active Comparator): Liraglutide: 3 mg/day sc. The GLP-1 RA, liraglutide (3.0 mg), or placebo, will be administrated once daily as subcutaneous injections in the abdomen or thigh. The starting dose is 0.6 mg with weekly increments of 0.6 mg until 3.0 mg is achieved. The titration procedure will be prolonged for participants who do not tolerate fast up-titration. Participants who do not tolerate the 3.0 mg dose may in special circumstances stay at lower dose (2.4 mg). However, the aim is to reach 3.0 mg for all study participants.
  Exercise: 150 min of moderate intensity, 75 min of vigorous intensity, or an equivalent combination of moderate and vigorous intensity exercise per week in accordance with WHO recommendations.
  Interventions: Drug: Liraglutide; Behavioral: Exercise
- Liraglutide + non-exercise (Other): Liraglutide: 3 mg/day sc. The GLP-1 RA, liraglutide (3.0 mg), or placebo, will be administrated once daily as subcutaneous injections in the abdomen or thigh. The starting dose is 0.6 mg with weekly increments of 0.6 mg until 3.0 mg is achieved. The titration procedure will be prolonged for participants who do not tolerate fast up-titration. Participants who do not tolerate the 3.0 mg dose may in special circumstances stay at lower dose (2.4 mg). However, the aim is to reach 3.0 mg for all study participants.
  Non-exercise: Participants should stay at same physical activity level (i.e. max. 2 h of vigorous endurance training/week) as when the participant was included in the study.
  Interventions: Drug: Liraglutide
- Placebo + exercise (Other): Placebo: 3mg/day sc.
  Exercise: 150 min of moderate intensity, 75 min of vigorous intensity, or an equivalent combination of moderate and vigorous intensity exercise per week in accordance with WHO recommendations.
  Interventions: Behavioral: Exercise
- Placebo + non-exercise (No Intervention): Placebo: 3mg/day sc.
  Non-exercise: Participants should stay at same physical activity level (i.e. max. 2 h of vigorous endurance training/week) as when the participant was included in the study.

INTERVENTIONS:
Drug: Liraglutide — Daily injections (3mg) with weight consultations starting at dose of 0.6 mg injections with 0.6 mg increments weekly until 3.0 mg is achieved. For subjects who do not tolerate the fast weekly up-titration of 0.6 mg study drug until the 3mg, the titration procedure can be prolonged with up to three weeks for each up-titration.
  Subjects who do not tolerate the 3mg dose may in special circumstances stay at 2.4 mg, however the overall aim is to reach 3 mg for all study subjects.
  The dosage and up-titration follow the recommendations from the summary of product characteristics.
  Other Names: Saxenda
  Arms: Liraglutide + exercise; Liraglutide + non-exercise
Behavioral: Exercise — 150 min of moderate intensity, 75 min of vigorous intensity, or an equivalent combination of moderate and vigorous intensity exercise per week in accordance with WHO recommendations.
  Exercise prescription will be performed under strict control of the scientific personnel.
  There will be aerobic exercise and will include 4 sessions per week after the ramp-in period.
  2 sessions per week will be performed under supervision of the staff and 2 sessions will be performed individually but monitored by the staff.
  Supervised sessions include structured exercise with a duration of 45 min. Of this 30 min will comprise of interval-based spinning session and 15 min circuit training program focusing on large muscle groups.
  Individual exercise includes aerobic exercise and general physical activity (e.g brisk walking and cycling to work).
  Participants will use heart rate monitors during sessions.
  Arms: Liraglutide + exercise; Placebo + exercise

SUMMARY:
Introduction: The success rate of weight loss maintenance is limited. Therefore, the purpose of this study is to investigate the maintenance of weight loss and immunometabolic health outcomes after diet-induced weight loss followed by one-year treatment with a glucagon-like peptide-1 receptor agonist (liraglutide), physical exercise, or the combination of both treatments as compared with placebo in individuals with obesity.

Methods and analysis: This is an investigator-initiated, randomized, placebo-controlled, parallel group trial. The investigators will enroll women and men (age 18 to 65 years) with obesity (body mass index 32 to 43 kg/m2) to adhere to a very low-calorie diet (800 kcal/day) for eight weeks in order to lose at least 5 % of body weight. Subsequently, participants will be randomized in a 1:1:1:1 ratio to one of four study groups for 52 weeks: 1) placebo, 2) exercise 150 min/week + placebo, 3) liraglutide 3.0 mg/day, and 4) exercise 150 min/week + liraglutide 3.0 mg/day. Re-screening is allowed within the recruitment period.

The primary endpoint is change in body weight from randomization to end-of-treatment.

Ethics and dissemination: The trial has been approved by the ethical committee of the Capital Region of Denmark (H-16027082) and the Danish Medicines Agency (EudraCT 2015-005585-32). The trial will be conducted in agreement with the Declaration of Helsinki and monitored to follow the guidelines for good clinical practice. Results will be submitted for publication in international peer-reviewed scientific journals.

DETAILED DESCRIPTION:
Obesity is associated with increased risk of developing cardiovascular disease and type 2 diabetes (T2D), along with increased risk of all-cause mortality [1,2]. Obesity management guidelines recommends weight loss of more than 5 % of initial body weight to improve cardiometabolic risk factors, with greater weight loss producing greater benefits [3,4]. A 5 to 10 % weight loss improves lipid profile (~20% reduction in triglycerides, ~15 % reduction in LDL-cholesterol, ~8 % increase in HDL-cholesterol levels) [1,4,5], reduces systolic and diastolic blood pressure (~5 and ~4 mmHg, respectively) [3,6], reduces HbA1c [3,4], and improves insulin sensitivity [7-9]. However, weight regain reverse these health benefits [10,11]. Furthermore, intentional weight loss is typically followed by a 30 to 50 % regain of lost weight within the first year [12-14]. The main biological reasons for the rapid weight regain may be that weight loss causes a decrease in total energy expenditure to a degree that is greater than predicted from the decrease in fat and lean mass [15,16] in combination with increased appetite in the weight-reduced state [17,18].

Increasing energy expenditure by increasing physical activity is the first-line lifestyle modification in the treatment of obesity along with reducing food intake. For exercise interventions targeting general public health recommendations (at least 150 min/week of moderate intensity aerobic exercise), the associated weight loss is often modest (0-3 %) without concomitant calorie restriction [19-21]. However, independent of weight loss, increasing physical activity improves body composition, glycemic control, low grade inflammatory profile, and cardiorespiratory fitness in individuals with overweight and obesity [22-25]. In addition, exercise may preserve lean mass during weight loss [26] and thereby counteract the associated decrease in resting metabolic rate [27], which may explain the observation that individuals performing regular exercise have less body weight regain after weight loss compared to participants that do not exercise [28,29].

Glucagon-like peptide-1 (GLP-1) is an incretin hormone primarily secreted from enteroendocrine L-cells in the gut after food intake. GLP-1 stimulates glucose-dependent insulin secretion thereby lowering blood glucose and reduces appetite and thereby food intake [30,31]. Treatment for 56 weeks with the GLP-1 receptor agonist (GLP-1 RA), liraglutide (3.0 mg), as an adjunct to regular diet and physical activity recommendations has been shown to improve glycemic control and induce moderate weight loss of 4.0 % in patients with T2D [32] and 5.4 % in non-diabetic individuals with overweight or obesity [33] compared to placebo. In addition, liraglutide has been shown to maintain a diet-induced weight loss over 56 weeks [34] and maintain very low-calorie diet-induced improvements of fasting plasma glucose and triglycerides over 52 weeks of weight loss maintenance superior to similar diet-induced weight loss maintenance in obese nondiabetic individuals [18].

Obesity is associated with chronic low-grade inflammation [35,36] which is linked to the development of atherosclerosis and insulin resistance [37-39]. Physically active individuals have lower inflammatory biomarker concentrations than their inactive counterparts [24], possibly explained by antiinflammatory effects of an acute bout of exercise [40] and lower levels of visceral adipose tissue [41]. GLP-1 has also emerged as an immunomodulatory agent [42,43]. In mice, GLP-1 RA administration reduces macrophage accumulation and inflammatory markers in the arterial wall [44], adipose tissue [45], and heart [46]. Similarly, GLP-1 RAs have shown antiinflammatory effects in human coronary artery endothelial cells and aortic endothelial cells [47]. In humans with T2D, short term GLP-1 RA treatment exert antiinflammatory actions, reflected in reduced levels of the macrophage activation molecule sCD163 [48] and reduced production of several proinflammatory markers, such as TNF-α, IL1β, and IL-6 in peripheral blood mononuclear cells [48,49]. Another study showed no improvement of obesity-associated adipose tissue dysfunction in T2D patients after GLP-1RA treatment [50]. One year treatment with GLP-1 RAs reduce the inflammation marker, high-sensitivity C-reactive protein, in overweight and obese individuals [33] and T2D patients [51]. Notably, in patients with T2D and high cardiovascular risk, GLP-1 RAs reduced the rate of occurrence of first major cardiovascular event [52,53].

Thus, both physical activity and GLP-1 RA treatment seem to facilitate weight loss maintenance, improve metabolic health, and reduce systemic inflammation. However, diet-induced weight loss decreases energy expenditure and increases appetite. The investigators hypothesize that the combination of physical activity and liraglutide treatment improves weight loss maintenance and immunometabolic health since the decreased energy expenditure is targeted with exercise and the increased appetite with liraglutide.

Objective:

The objectives of this study are to investigate the maintenance of weight loss and immunometabolic health outcomes over 52 weeks with liraglutide treatment, physical exercise, and the combination in individuals with obesity, after a very low-calorie diet.

Endpoints:

Primary endpoint: The primary endpoint is change in body weight from after the initial weight loss phase (baseline/V1) to end of treatment after 52 weeks (end/V3).

Secondary endpoints: The secondary endpoints are changes in a) body composition (fat %, lean and fat mass ) and b) metabolic health (glucose tolerance (HOMA-IR, Matsuda, HbA1c), lipid status, waist circumference, blood pressure) from V1 to V3.

Other prespecified endpoints:

Prespecified endpoints include changes from V0 to V1 to V3 in the following parameters:

* Physical fitness (measured by VO2 peak test on a bike, strength test, and functional stair test)
* Fasting and meal-related hormonal response (e.g. GLP-1, PYY, ghrelin, leptin, etc.)
* Food preferences and subjective appetite sensation (measured by the Leeds Food Preference Questionnaire (LFPQ) and visual analogue scales)
* Determination of daily physical activity and sleep (measured by triaxial accelerometry (GENEActiv, ActivInsights Ltd, UK) and questionnaires (PSQI and IPAQ)).
* Endothelial function (e.g. measured by flow-mediated dilation (FMD) and relevant systemic biomarkers)
* Standard clinical blood samples (e.g. C-reactive protein, vitamin D, and glycated hemoglobin)
* Electrocardiogram (ECG)
* Heart rate
* Health-related questionnaires (self-rated quality of life (The Short Form (36) Health Survey), eating habits (three-factor eating questionnaire), physical activity (International Physical Activity Questionnaire), sleep quality (Pittsburgh Sleep Quality Index), and self-efficacy (General Self-Efficacy Scale).
* Systemic markers of immunometabolism (e.g. measured by single cell analysis)
* Immunometabolic changes in the subcutaneous adipose tissue (e.g. measured by single cell analysis)
* Gene expression profile of circulating inflammatory cells (e.g. in adipose tissue cells in which proinflammatory and antiinflammatory adipocytokines, adipocyte differentiation markers, and markers of macrophages infiltration will be determined by reverse transcription-qPCR).
* Bone health (measured by DXA scan and relevant systemic bone markers)
* Faecal bacterial composition
* Metabolomics and proteomics
* Epigenetics of spermatozoa
* Use of medication
* Proportion of participants with 5,10, 15 and 20% total weight loss
* Weight loss from V0-V3

Follow-up visit 1 year after end of treatment:

* Body weight, height, waist and hip circumference, blood pressure and pulse
* Fasting blood samples (identical to samples obtained for V0)
* DEXA scan
* Questionnaires as in V0
* Accelerometer device (GENEActiv) worn on wrist for 7 consecutive days and nights after follow-up testing to assess physical activity levels

ELIGIBILITY:
Inclusion Criteria:

* BMI > 32 and < 43 (kg/m2)
* Age >18 and <65 years
* Safe contraceptive method

Exclusion Criteria:

* Patients diagnosed with known serious chronic illness including type 1 or 2 diabetes (or a randomly measured fasting plasma glucose > 7 mmol/l)
* Angina pectoris, coronary heart disease, congestive heart failure (NYHA III-IV)
* Severe renal impairment (creatinine clearance (GFR) <30 mL/min)
* Severe hepatic impairment
* Inflammatory bowel disease
* Gastroparesis
* Cancer
* Chronic obstructive lung disease
* Psychiatric disease, a history of major depressive or other severe psychiatric disorders
* The use of medications that cause clinically significant weight gain or loss
* Previous bariatric surgery
* A history of idiopathic acute pancreatitis
* A family or personal history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma
* Osteoarthritis which is judged to be too severe to manage the exercise programme. As intended per study design the intervention will include a 5% weight loss prior to randomization, thus it is expected that possible participants with mild form of osteoarthritis will be able to manage exercise prescriptions.
* Pregnancy, expecting pregnancy or breast feeding. If a study participant is in doubt whether she could be pregnant, a urine pregnancy test is performed. Females of childbearing potential who are not using adequate contraceptive methods (as required by local law or practice). Adequate contraception must be used throughout the study period and at least 65 hours after discontinuation of trial medication (65 hours corresponds to 5 times the half-life of Saxenda). Allergy to any of the ingredients/excipients.
* Allergy to any of the ingredients/excipients of the study medication: liraglutide, disodium phosphate dihydrate, propylene glycol, phenol, hydrochloric acid, sodium hydroxide.
* Regular exercise training at high intensity (e.g. spinning) >2 hours per week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Body weight change (kg) | Change from baseline to end-of-treatment (52 weeks)
  Weight will be measured to the nearest 0.1 kg. The same set of scales should ideally be used throughout the trial. Weight should be measured in a fasting state without shoes and wearing light clothes.

SECONDARY OUTCOMES:
Body composition (fat percentage) | Change from baseline to end-of-treatment (52 weeks)
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure body fat percentage (%).
Body composition (fat mass and fat free mass) | Change from baseline to end-of-treatment (52 weeks)
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure fat mass/fat free mass (kg).
Waist and hip circumference | Change from baseline to end-of-treatment (52 weeks)
  Waist circumference, the midpoint between lowest rib and iliac crest, and hip circumference, the level of the great trochanters, will be measured in duplicate to the nearest 0.1 cm after gentle expiration.
HOMA-IR | Change from baseline to end-of-treatment (52 weeks)
  Fasting insulin (μU/mL) * fasting glucose (mmol/L) / 22.5
Matsuda Index | Change from baseline to end-of-treatment (52 weeks)
  10000/sqrt(fasting glucose * fasting insulin * mean glucose * mean insulin)
Hormonal regulation of blood glucose | Change from baseline to end-of-treatment (52 weeks)
  Measured from blood samples (e.g. glucose tolerance, HbA1c (mmol/mol))
Lipids | Change from baseline to end-of-treatment (52 weeks)
  Measured from blood samples (e.g. cholesterol (HDL, LDL, VLDL) and triglycerides (TG)) (mmol/L)
Blood pressure | Change from baseline to end-of-treatment (52 weeks)
  Blood pressure (systolic/diastolic) will be measured in duplicate from the non-dominant arm with a digital blood pressure monitor in sitting position after at least 5 min of rest (mmHg).
Metabolic Syndrome (yes/no) | Change from baseline to end-of-treatment (52 weeks)
  Relevant clinical parameters lipids, fasting glucose, waist circumference, and blood pressure will be used to investigate whether the participants have metabolic syndrome (unit: yes/no).
MetS (z-score) | Change from baseline to end-of-treatment (52 weeks)
  Relevant clinical parameters lipids, fasting glucose, waist circumference, and blood pressure will be used to calculate a z-score (unit: z-score)

OTHER OUTCOMES:
Physical fitness (ml/min/min) | Change from baseline to end-of-treatment (52 weeks)
  Measured by VO2 peak test on a bike, strength test, and functional stair test (unit: ml/min/min)
Quality of life score | Change from baseline to end-of-treatment (52 weeks)
  The Short Form 36 Health Survey, (units on a scale: 0-100). Higher scores mean a better outocome
Heart rate | Change from screening to baseline to end-of-treatment (52 weeks)
  Heart rate (bpm)
Proportion of participants with % weight loss | Change from screening to end-of-treatment (52 weeks)
  Proportion of participants with % weight loss (%)
Total weight loss | Change from screening to end-of-treatment (52 weeks)
  Total weight loss (%)
Questionnaires | Change from baseline to end-of-treatment (52 weeks)
  Scores (units on a scale)
Fasting and meal-related hormonal response | Change from baseline to end-of-treatment (52 weeks)
  Blood samples
Food preferences/subjective appetite sensation | Change from baseline to end-of-treatment (52 weeks)
  Scores
Endothelial function | Change from screening to baseline to end-of-treatment (52 weeks)
  Measured by flow-mediated dilation (%)
Determination of daily physical activity/sleep | Change from screening to baseline to end-of-treatment (52 weeks)
  Measured by triaxial accelerometry (GENEActiv, ActivInsights Ltd, UK) (min/day).
Bone health (Bone mineral density) | Change from baseline to end-of-treatment (52 weeks)
  Measured by DXA scan (g/cm^2)
Systemic markers of immunometabolism | Change from screening to baseline to end-of-treatment (52 weeks)
  Immunometabolic composition (CRP mg/l)
Immunometabolic changes in the subcutaneous adipose tissue | Change from screening to baseline to end-of-treatment (52 weeks)
  Immunometabolic composition (gene expression)
Spermatozoa | Change from screening to baseline to end-of-treatment (52 weeks)
  Spermatozoa concentration (counts/ml)
Faecal bacterial composition | Change from screening to baseline to end-of-treatment (52 weeks)
  Microbiome composition
Use of medication | Change from screening to baseline to end-of-treatment (52 weeks)
  n, frequency
Follow-up visit | End-of-treatment to 1 year after intervention
  one-year follow-up (kg/fat%)

CONTACTS AND LOCATIONS:
Overall Officials: Signe S Torekov, Prof, PhD, Study Director — University of Copenhagen; Sten Madsbad, Prof, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

REFERENCES:
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Abdelaal M, le Roux CW, Docherty NG. Morbidity and mortality associated with obesity. Ann Transl Med. 2017 Apr;5(7):161. doi: 10.21037/atm.2017.03.107. PMID 28480197
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITY. Endocr Pract. 2016 Jul;22 Suppl 3:1-203. doi: 10.4158/EP161365.GL. Epub 2016 May 24. PMID 27219496
- [Background] Nordmann AJ, Nordmann A, Briel M, Keller U, Yancy WS Jr, Brehm BJ, Bucher HC. Effects of low-carbohydrate vs low-fat diets on weight loss and cardiovascular risk factors: a meta-analysis of randomized controlled trials. Arch Intern Med. 2006 Feb 13;166(3):285-93. doi: 10.1001/archinte.166.3.285. PMID 16476868
- [Background] Weiss EP, Albert SG, Reeds DN, Kress KS, McDaniel JL, Klein S, Villareal DT. Effects of matched weight loss from calorie restriction, exercise, or both on cardiovascular disease risk factors: a randomized intervention trial. Am J Clin Nutr. 2016 Sep;104(3):576-86. doi: 10.3945/ajcn.116.131391. Epub 2016 Jul 27. PMID 27465384
- [Background] Weiss EP, Reeds DN, Ezekiel UR, Albert SG, Villareal DT. Circulating cytokines as determinants of weight loss-induced improvements in insulin sensitivity. Endocrine. 2017 Jan;55(1):153-164. doi: 10.1007/s12020-016-1093-4. Epub 2016 Sep 7. PMID 27605038
- [Background] Magkos F, Fraterrigo G, Yoshino J, Luecking C, Kirbach K, Kelly SC, de las Fuentes L, He S, Okunade AL, Patterson BW, Klein S. Effects of Moderate and Subsequent Progressive Weight Loss on Metabolic Function and Adipose Tissue Biology in Humans with Obesity. Cell Metab. 2016 Apr 12;23(4):591-601. doi: 10.1016/j.cmet.2016.02.005. Epub 2016 Feb 22. PMID 26916363
- [Background] Trussardi Fayh AP, Lopes AL, Fernandes PR, Reischak-Oliveira A, Friedman R. Impact of weight loss with or without exercise on abdominal fat and insulin resistance in obese individuals: a randomised clinical trial. Br J Nutr. 2013 Aug 28;110(3):486-92. doi: 10.1017/S0007114512005442. Epub 2013 Jan 10. PMID 23302544
- [Background] Kroeger CM, Hoddy KK, Varady KA. Impact of weight regain on metabolic disease risk: a review of human trials. J Obes. 2014;2014:614519. doi: 10.1155/2014/614519. Epub 2014 Aug 14. PMID 25197563
- [Background] Thomas TR, Warner SO, Dellsperger KC, Hinton PS, Whaley-Connell AT, Rector RS, Liu Y, Linden MA, Chockalingam A, Thyfault JP, Huyette DR, Wang Z, Cox RH. Exercise and the metabolic syndrome with weight regain. J Appl Physiol (1985). 2010 Jul;109(1):3-10. doi: 10.1152/japplphysiol.01361.2009. Epub 2010 Feb 18. PMID 20167668
- [Background] Barte JC, ter Bogt NC, Bogers RP, Teixeira PJ, Blissmer B, Mori TA, Bemelmans WJ. Maintenance of weight loss after lifestyle interventions for overweight and obesity, a systematic review. Obes Rev. 2010 Dec;11(12):899-906. doi: 10.1111/j.1467-789X.2010.00740.x. PMID 20345430
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Curioni CC, Lourenco PM. Long-term weight loss after diet and exercise: a systematic review. Int J Obes (Lond). 2005 Oct;29(10):1168-74. doi: 10.1038/sj.ijo.0803015. PMID 15925949
- [Background] Rosenbaum M, Leibel RL. Adaptive thermogenesis in humans. Int J Obes (Lond). 2010 Oct;34 Suppl 1(0 1):S47-55. doi: 10.1038/ijo.2010.184. PMID 20935667
- [Background] Leibel RL, Rosenbaum M, Hirsch J. Changes in energy expenditure resulting from altered body weight. N Engl J Med. 1995 Mar 9;332(10):621-8. doi: 10.1056/NEJM199503093321001. PMID 7632212
- [Background] Iepsen EW, Lundgren J, Holst JJ, Madsbad S, Torekov SS. Successful weight loss maintenance includes long-term increased meal responses of GLP-1 and PYY3-36. Eur J Endocrinol. 2016 Jun;174(6):775-84. doi: 10.1530/EJE-15-1116. Epub 2016 Mar 14. PMID 26976129
- [Background] Iepsen EW, Lundgren J, Dirksen C, Jensen JE, Pedersen O, Hansen T, Madsbad S, Holst JJ, Torekov SS. Treatment with a GLP-1 receptor agonist diminishes the decrease in free plasma leptin during maintenance of weight loss. Int J Obes (Lond). 2015 May;39(5):834-41. doi: 10.1038/ijo.2014.177. Epub 2014 Oct 7. PMID 25287751
- [Background] Swift DL, Johannsen NM, Lavie CJ, Earnest CP, Church TS. The role of exercise and physical activity in weight loss and maintenance. Prog Cardiovasc Dis. 2014 Jan-Feb;56(4):441-7. doi: 10.1016/j.pcad.2013.09.012. Epub 2013 Oct 11. PMID 24438736
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Shaw K, Gennat H, O'Rourke P, Del Mar C. Exercise for overweight or obesity. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD003817. doi: 10.1002/14651858.CD003817.pub3. PMID 17054187
- [Background] Nordby P, Auerbach PL, Rosenkilde M, Kristiansen L, Thomasen JR, Rygaard L, Groth R, Brandt N, Helge JW, Richter EA, Ploug T, Stallknecht B. Endurance training per se increases metabolic health in young, moderately overweight men. Obesity (Silver Spring). 2012 Nov;20(11):2202-12. doi: 10.1038/oby.2012.70. Epub 2012 Mar 22. PMID 22436841
- [Background] Bruce CR, Thrush AB, Mertz VA, Bezaire V, Chabowski A, Heigenhauser GJ, Dyck DJ. Endurance training in obese humans improves glucose tolerance and mitochondrial fatty acid oxidation and alters muscle lipid content. Am J Physiol Endocrinol Metab. 2006 Jul;291(1):E99-E107. doi: 10.1152/ajpendo.00587.2005. Epub 2006 Feb 7. PMID 16464906
- [Background] You T, Arsenis NC, Disanzo BL, Lamonte MJ. Effects of exercise training on chronic inflammation in obesity : current evidence and potential mechanisms. Sports Med. 2013 Apr;43(4):243-56. doi: 10.1007/s40279-013-0023-3. PMID 23494259
- [Background] Lavie CJ, Arena R, Swift DL, Johannsen NM, Sui X, Lee DC, Earnest CP, Church TS, O'Keefe JH, Milani RV, Blair SN. Exercise and the cardiovascular system: clinical science and cardiovascular outcomes. Circ Res. 2015 Jul 3;117(2):207-19. doi: 10.1161/CIRCRESAHA.117.305205. PMID 26139859
- [Background] Calbet JAL, Ponce-Gonzalez JG, Calle-Herrero J, Perez-Suarez I, Martin-Rincon M, Santana A, Morales-Alamo D, Holmberg HC. Exercise Preserves Lean Mass and Performance during Severe Energy Deficit: The Role of Exercise Volume and Dietary Protein Content. Front Physiol. 2017 Jul 24;8:483. doi: 10.3389/fphys.2017.00483. eCollection 2017. PMID 28790922
- [Background] Stiegler P, Cunliffe A. The role of diet and exercise for the maintenance of fat-free mass and resting metabolic rate during weight loss. Sports Med. 2006;36(3):239-62. doi: 10.2165/00007256-200636030-00005. PMID 16526835
- [Background] Jakicic JM, Marcus BH, Lang W, Janney C. Effect of exercise on 24-month weight loss maintenance in overweight women. Arch Intern Med. 2008 Jul 28;168(14):1550-9; discussion 1559-60. doi: 10.1001/archinte.168.14.1550. PMID 18663167
- [Background] Wing RR, Phelan S. Long-term weight loss maintenance. Am J Clin Nutr. 2005 Jul;82(1 Suppl):222S-225S. doi: 10.1093/ajcn/82.1.222S. PMID 16002825
- [Background] Flint A, Raben A, Astrup A, Holst JJ. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998 Feb 1;101(3):515-20. doi: 10.1172/JCI990. PMID 9449682
- [Background] Holst JJ, Deacon CF, Vilsboll T, Krarup T, Madsbad S. Glucagon-like peptide-1, glucose homeostasis and diabetes. Trends Mol Med. 2008 Apr;14(4):161-8. doi: 10.1016/j.molmed.2008.01.003. Epub 2008 Mar 18. PMID 18353723
- [Background] Davies MJ, Bergenstal R, Bode B, Kushner RF, Lewin A, Skjoth TV, Andreasen AH, Jensen CB, DeFronzo RA; NN8022-1922 Study Group. Efficacy of Liraglutide for Weight Loss Among Patients With Type 2 Diabetes: The SCALE Diabetes Randomized Clinical Trial. JAMA. 2015 Aug 18;314(7):687-99. doi: 10.1001/jama.2015.9676. PMID 26284720
- [Background] Pi-Sunyer X, Astrup A, Fujioka K, Greenway F, Halpern A, Krempf M, Lau DC, le Roux CW, Violante Ortiz R, Jensen CB, Wilding JP; SCALE Obesity and Prediabetes NN8022-1839 Study Group. A Randomized, Controlled Trial of 3.0 mg of Liraglutide in Weight Management. N Engl J Med. 2015 Jul 2;373(1):11-22. doi: 10.1056/NEJMoa1411892. PMID 26132939
- [Background] Wadden TA, Hollander P, Klein S, Niswender K, Woo V, Hale PM, Aronne L; NN8022-1923 Investigators. Weight maintenance and additional weight loss with liraglutide after low-calorie-diet-induced weight loss: the SCALE Maintenance randomized study. Int J Obes (Lond). 2013 Nov;37(11):1443-51. doi: 10.1038/ijo.2013.120. Epub 2013 Jul 1. PMID 23812094
- [Background] Stepien M, Stepien A, Wlazel RN, Paradowski M, Banach M, Rysz J. Obesity indices and inflammatory markers in obese non-diabetic normo- and hypertensive patients: a comparative pilot study. Lipids Health Dis. 2014 Feb 8;13:29. doi: 10.1186/1476-511X-13-29. PMID 24507240
- [Background] Panagiotakos DB, Pitsavos C, Yannakoulia M, Chrysohoou C, Stefanadis C. The implication of obesity and central fat on markers of chronic inflammation: The ATTICA study. Atherosclerosis. 2005 Dec;183(2):308-15. doi: 10.1016/j.atherosclerosis.2005.03.010. Epub 2005 Apr 25. PMID 16285994
- [Background] Duncan BB, Schmidt MI, Pankow JS, Ballantyne CM, Couper D, Vigo A, Hoogeveen R, Folsom AR, Heiss G; Atherosclerosis Risk in Communities Study. Low-grade systemic inflammation and the development of type 2 diabetes: the atherosclerosis risk in communities study. Diabetes. 2003 Jul;52(7):1799-805. doi: 10.2337/diabetes.52.7.1799. PMID 12829649
- [Background] Vozarova B, Weyer C, Lindsay RS, Pratley RE, Bogardus C, Tataranni PA. High white blood cell count is associated with a worsening of insulin sensitivity and predicts the development of type 2 diabetes. Diabetes. 2002 Feb;51(2):455-61. doi: 10.2337/diabetes.51.2.455. PMID 11812755
- [Background] Starkie R, Ostrowski SR, Jauffred S, Febbraio M, Pedersen BK. Exercise and IL-6 infusion inhibit endotoxin-induced TNF-alpha production in humans. FASEB J. 2003 May;17(8):884-6. doi: 10.1096/fj.02-0670fje. Epub 2003 Mar 5. PMID 12626436
- [Background] Gleeson M, Bishop NC, Stensel DJ, Lindley MR, Mastana SS, Nimmo MA. The anti-inflammatory effects of exercise: mechanisms and implications for the prevention and treatment of disease. Nat Rev Immunol. 2011 Aug 5;11(9):607-15. doi: 10.1038/nri3041. PMID 21818123
- [Background] Torekov SS. Glucagon-like peptide-1 receptor agonists and cardiovascular disease: from LEADER to EXSCEL. Cardiovasc Res. 2018 Aug 1;114(10):e70-e71. doi: 10.1093/cvr/cvy124. No abstract available. PMID 30052921
- [Background] Insuela DBR, Carvalho VF. Glucagon and glucagon-like peptide-1 as novel anti-inflammatory and immunomodulatory compounds. Eur J Pharmacol. 2017 Oct 5;812:64-72. doi: 10.1016/j.ejphar.2017.07.015. Epub 2017 Jul 6. PMID 28688914
- [Background] Arakawa M, Mita T, Azuma K, Ebato C, Goto H, Nomiyama T, Fujitani Y, Hirose T, Kawamori R, Watada H. Inhibition of monocyte adhesion to endothelial cells and attenuation of atherosclerotic lesion by a glucagon-like peptide-1 receptor agonist, exendin-4. Diabetes. 2010 Apr;59(4):1030-7. doi: 10.2337/db09-1694. Epub 2010 Jan 12. PMID 20068138
- [Background] Lee YS, Park MS, Choung JS, Kim SS, Oh HH, Choi CS, Ha SY, Kang Y, Kim Y, Jun HS. Glucagon-like peptide-1 inhibits adipose tissue macrophage infiltration and inflammation in an obese mouse model of diabetes. Diabetologia. 2012 Sep;55(9):2456-68. doi: 10.1007/s00125-012-2592-3. Epub 2012 Jun 22. PMID 22722451
- [Background] Noyan-Ashraf MH, Shikatani EA, Schuiki I, Mukovozov I, Wu J, Li RK, Volchuk A, Robinson LA, Billia F, Drucker DJ, Husain M. A glucagon-like peptide-1 analog reverses the molecular pathology and cardiac dysfunction of a mouse model of obesity. Circulation. 2013 Jan 1;127(1):74-85. doi: 10.1161/CIRCULATIONAHA.112.091215. Epub 2012 Nov 27. PMID 23186644
- [Background] Garczorz W, Gallego-Colon E, Kosowska A, Klych-Ratuszny A, Wozniak M, Marcol W, Niesner KJ, Francuz T. Exenatide exhibits anti-inflammatory properties and modulates endothelial response to tumor necrosis factor alpha-mediated activation. Cardiovasc Ther. 2018 Apr;36(2). doi: 10.1111/1755-5922.12317. Epub 2018 Jan 24. PMID 29283509
- [Background] Hogan AE, Gaoatswe G, Lynch L, Corrigan MA, Woods C, O'Connell J, O'Shea D. Glucagon-like peptide 1 analogue therapy directly modulates innate immune-mediated inflammation in individuals with type 2 diabetes mellitus. Diabetologia. 2014 Apr;57(4):781-4. doi: 10.1007/s00125-013-3145-0. Epub 2013 Dec 21. PMID 24362727
- [Background] Chaudhuri A, Ghanim H, Vora M, Sia CL, Korzeniewski K, Dhindsa S, Makdissi A, Dandona P. Exenatide exerts a potent antiinflammatory effect. J Clin Endocrinol Metab. 2012 Jan;97(1):198-207. doi: 10.1210/jc.2011-1508. Epub 2011 Oct 19. PMID 22013105
- [Background] Pastel E, McCulloch LJ, Ward R, Joshi S, Gooding KM, Shore AC, Kos K. GLP-1 analogue-induced weight loss does not improve obesity-induced AT dysfunction. Clin Sci (Lond). 2017 Mar 1;131(5):343-353. doi: 10.1042/CS20160803. Epub 2017 Jan 3. PMID 28049736
- [Background] Bunck MC, Diamant M, Eliasson B, Corner A, Shaginian RM, Heine RJ, Taskinen MR, Yki-Jarvinen H, Smith U. Exenatide affects circulating cardiovascular risk biomarkers independently of changes in body composition. Diabetes Care. 2010 Aug;33(8):1734-7. doi: 10.2337/dc09-2361. Epub 2010 Apr 27. PMID 20424219
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Derived] Jensen SBK, Fiorenza M, Juhl CR, Sandsdal RM, Jensen E, Seier SS, Janus C, Jorgensen JR, Blond MB, Holst JJ, Stallknecht BM, Madsbad S, Bandholm T, Torekov SS. Physical Fitness with Exercise and GLP-1 Receptor Agonist Treatment Alone or Combined After Diet-Induced Weight Loss: A Secondary Analysis of a Randomized Controlled Trial in Adults with Obesity. Sports Med. 2026 Jan 24. doi: 10.1007/s40279-025-02386-0. Online ahead of print. PMID 41579235
- [Derived] Holt J, Sandsdal RM, Byberg S, Janus C, Juhl CR, Jorgensen JR, Hartmann B, Stallknecht B, Holst JJ, Madsbad S, Jensen SBK, Torekov SS. One Year of Exercise After Weight Loss Increases Postprandial GLP-1 Secretion in Contrast to Usual Activity or GLP-1 Receptor Agonist Treatment. Obesity (Silver Spring). 2026 Jan;34(1):51-57. doi: 10.1002/oby.70043. Epub 2025 Sep 25. PMID 40998556
- [Derived] Holt R, Holt J, Jorsal MJ, Sandsdal RM, Jensen SBK, Byberg S, Juhl CR, Lundgren JR, Janus C, Stallknecht BM, Holst JJ, Juul A, Madsbad S, Jensen MB, Torekov SS. Weight Loss Induces Changes in Vitamin D Status in Women With Obesity But Not in Men: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2025 Jul 15;110(8):2215-2224. doi: 10.1210/clinem/dgae775. PMID 39530599
- [Derived] Jensen SBK, Blond MB, Sandsdal RM, Olsen LM, Juhl CR, Lundgren JR, Janus C, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Healthy weight loss maintenance with exercise, GLP-1 receptor agonist, or both combined followed by one year without treatment: a post-treatment analysis of a randomised placebo-controlled trial. EClinicalMedicine. 2024 Feb 19;69:102475. doi: 10.1016/j.eclinm.2024.102475. eCollection 2024 Mar. PMID 38544798
- [Derived] Sandsdal RM, Juhl CR, Jensen SBK, Lundgren JR, Janus C, Blond MB, Rosenkilde M, Bogh AF, Gliemann L, Jensen JB, Antoniades C, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Combination of exercise and GLP-1 receptor agonist treatment reduces severity of metabolic syndrome, abdominal obesity, and inflammation: a randomized controlled trial. Cardiovasc Diabetol. 2023 Feb 25;22(1):41. doi: 10.1186/s12933-023-01765-z. PMID 36841762
- [Derived] Bogh AF, Jensen SBK, Juhl CR, Janus C, Sandsdal RM, Lundgren JR, Noer MH, Vu NQ, Fiorenza M, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Insufficient sleep predicts poor weight loss maintenance after 1 year. Sleep. 2023 May 10;46(5):zsac295. doi: 10.1093/sleep/zsac295. PMID 36472579
- [Derived] Jensen SBK, Janus C, Lundgren JR, Juhl CR, Sandsdal RM, Olsen LM, Andresen A, Borg SA, Jacobsen IC, Finlayson G, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Exploratory analysis of eating- and physical activity-related outcomes from a randomized controlled trial for weight loss maintenance with exercise and liraglutide single or combination treatment. Nat Commun. 2022 Aug 15;13(1):4770. doi: 10.1038/s41467-022-32307-y. PMID 35970829
- [Derived] Andersen E, Juhl CR, Kjoller ET, Lundgren JR, Janus C, Dehestani Y, Saupstad M, Ingerslev LR, Duun OM, Jensen SBK, Holst JJ, Stallknecht BM, Madsbad S, Torekov SS, Barres R. Sperm count is increased by diet-induced weight loss and maintained by exercise or GLP-1 analogue treatment: a randomized controlled trial. Hum Reprod. 2022 Jun 30;37(7):1414-1422. doi: 10.1093/humrep/deac096. PMID 35580859
- [Derived] Lundgren JR, Janus C, Jensen SBK, Juhl CR, Olsen LM, Christensen RM, Svane MS, Bandholm T, Bojsen-Moller KN, Blond MB, Jensen JB, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Healthy Weight Loss Maintenance with Exercise, Liraglutide, or Both Combined. N Engl J Med. 2021 May 6;384(18):1719-1730. doi: 10.1056/NEJMoa2028198. PMID 33951361

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT04122716/SAP_001.pdf